CLINICAL TRIAL: NCT04628806
Title: Heat Shock Protein (HSP) 70 to Quantify and Characterize Circulating Tumor Cells in Patients With Advanced or Metastatic Tumors.
Brief Title: Heat Shock Protein (HSP) 70 to Quantify and Characterize Circulating Tumor Cells
Acronym: HSP70CTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Klinikum rechts der Isar, TU München, (TUM), Munich, Germany. (Unknown)
Responsible Party: Principal Investigator, Sebastian Zschaeck, Doctor Sebastian Zschaeck, principal investigator, Charite University, Berlin, Germany
Other Study IDs: HSP70CTC
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Melanoma Stage IV; Sarcoma; Squamous Cell Carcinoma; Pancreatic Cancer Stage IV; Prostate Cancer; Breast Cancer Stage IV
MeSH Terms: conditions — Melanoma; Sarcoma; Carcinoma, Squamous Cell; Pancreatic Neoplasms; Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — circulating tumor cells and biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSP70CTC: Isolation of circulating tumor cells by HSP70
  Interventions: Diagnostic Test: CTC isolation by HSP70

INTERVENTIONS:
Diagnostic Test: CTC isolation by HSP70 — patients will receive additional blood examinations with quantification of circulating tumor cells by HSP70 antibodies and EpCAM.

SUMMARY:
This study investigates the ability of heat shock protein HSP70 to isolate and quantify circulating tumor cells (CTCs) in patients with advanced or metastatic tumors.

CTCs will be isolated from peripheral blood before antineoplastic treatment and again after three months. Isolation using HSP70 will be compared with standard CTC isolation by EpCAM.

Additionally, imaging parameters of the primary tumor (if available) and metastases will be analysed and correlations between molecular alterations and imaging parameters will be assesed.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic malignant melanoma (stage IV)
* Metastatic or unresectable pancreatic adenocarcinoma (stage III or IV)
* Metastatic breast cancer
* Metastatic sarcoma
* Metastatic squamous cell carcinoma of the cervix uteri, head and neck region, vulva, anus or penis
* hormone-refractory prostate cancer

Exclusion Criteria:

* psychiatric disorders that impede adequate informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oncological patients treated at a tertiary center
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Radiographic response to initial treatment | 3 months after study enrollment
  radiographic response to treatment will be scored according to RECIST criteria and associated with the number of CTC

SECONDARY OUTCOMES:
Correlation between number of CTC isolated with HSP70 compared to EpCAM | 3 months (at both CTC assessment timepoints)
  the number of CTCs obtained by the novel HSP70 method will be compared to the current gold standard that uses EpCAM. This will be performed for the whole cohort and separate for each tumor site
Correlation between differential expressed radiommic parameters between primary tumor and metastases and genetic alterations of the primary tumor and CTCs | 3 months (at both CTC assessment timepoints)
  computed tomography parameters of primary tumors and metastases will be analysed and parameters extraced that are differentially expressed between both. The same will be performed for genomic mutations and gene expression of the primary tumor and CTC. Correlation analyses will be performed to analyze if radiographic parameters resemble genetic alterations
Progression free survival | 2 years
  Progression free survival will be evaluated with the number of CTC as variable. This will be performed for the whole cohort and separate for each tumor site
Overall survival | 2 years
  Overall survival will be evaluated with the number of CTC as variable. This will be performed for the whole cohort and separate for each tumor site

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Zschaeck, MD, Principal Investigator — Charité
Locations (1):
- Klinik für Radioonkologie und Strahlentherapie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
patients can sign an optional agreement that their pseudonymized imaging and genetic data will be shared on cancerimagingarchive.net
Time Frame: data will be uploaded 2 years after study completion
Access Criteria: no specific criteria except proper referencing.
URL: https://www.cancerimagingarchive.net/

REFERENCES:
- [Derived] Roy AA, Pandey A, Dhas N, Hegde MM, Parekh HS, Andugulapati SB, Nandakumar K, Satish Rao BS, Mutalik S. The Confluence of Nanotechnology and Heat Shock Protein 70 in Pioneering Glioblastoma Multiforme Therapy: Forging Pathways Towards Precision Targeting and Transformation. Adv Pharmacol Pharm Sci. 2025 Apr 24;2025:1847197. doi: 10.1155/adpp/1847197. eCollection 2025. PMID 40313865